CLINICAL TRIAL: NCT05757713
Title: Single Arm, Open-label Study to Assess the Safety and Pharmacokinetics of a 14-day Regimen of Teplizumab in Pediatric Stage 2 Type 1 Diabetes (Participants <8 Years of Age With at Least Two Autoantibodies and Dysglycemia)
Brief Title: Teplizumab in Pediatric Stage 2 Type 1 Diabetes
Acronym: PETITE-T1D
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRV-031-005; SFY18116 (Other: Sanofi Identifier)
Record Dates: First submitted 2023-02-13; First posted 2023-03-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; Stage 2; Pediatric type 1 diabetes; T1D; At-risk
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Intervention Model Description: Single arm, non-randomized, open-label, multi-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- teplizumab injection (Experimental): teplizumab injection, sterile solution for intravenous use
  Interventions: Biological: teplizumab

INTERVENTIONS:
Biological: teplizumab — CD3-directed humanized monoclonal antibody

SUMMARY:
The purpose of this study is to assess the safety and pharmacokinetics (PK) of teplizumab in participants with Stage 2 type 1 diabetes who are <8 years of age.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized, open-label, multicenter study in the U.S. to assess the safety and pharmacokinetics of teplizumab in pediatric participants with Stage 2 type 1 diabetes (T1D) (two T1D-related autoantibodies and dysglycemia) who are 0 to <8 years of age. Anti-drug antibodies/neutralizing antibodies (ADA/NAb) will also be assessed.

Approximately 20 participants will be enrolled. The regimen consists of an intravenous infusion of teplizumab once daily for 14 consecutive days. The study duration for each individual may last up to approximately 26 months.

The safety, tolerability, PK, ADA, and T1D clinical feature data will be summarized using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a male or female 0 to < 8 years of age, inclusive, at Day 1
2. Participant has Stage 2 T1D (two T1D-related autoantibodies and dysglycemia)

Exclusion Criteria:

1. Participant has any autoimmune disease other than T1D with the exception of stable thyroid or celiac disease
2. Has an active infection and/or fever
3. Has a history of or serologic evidence at screening of current or past infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
4. Has any condition that, in the opinion of the Investigator, would interfere with the study conduct or the safety of the participant.

Ages: 0 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), TEAEs leading to withdrawal, and serious adverse events (SAEs) | Through 104 Weeks
  Safety and tolerability endpoint

SECONDARY OUTCOMES:
Serum concentrations of teplizumab | Sparse PK samples between Days 1 and 28
  Pharmacokinetic (PK) endpoint
Anti-drug antibody (ADA) titers and presence of neutralizing antibodies (Nab) | Through 104 weeks
  Immunogenicity endpoint
CD3 receptor occupancy | Days 1 and 9
  To assess the effects of teplizumab on cluster of differentiation 3 (CD3) receptor occupancy

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- United States (10):
  - UCSF Medical Center Site Number : 107, San Francisco, California
  - Barbara Davis Center for Diabetes Site Number : 102, Aurora, Colorado
  - Yale University School of Medicine Site Number : 101, New Haven, Connecticut
  - Centricity Research Site Number : 104, Columbus, Georgia
  - Indianapolis University Health Riley Hospital for Children Site Number : 110, Indianapolis, Indiana
  - UBMD Pediactrics Site Number : 105, Buffalo, New York
  - Children's Hospital of Philadelphia Site Number : 108, Philadelphia, Pennsylvania
  - Sanford Diabetes and Thyroid Clinic Site Number : 106, Sioux Falls, South Dakota
  - Vanderbilt Univerity Medical Center Site Number : 109, Nashville, Tennessee
  - MulitCare Institute for Research & Innovation Site Number : 103, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Gitelman SE, Simmons K, Sherr JL, Leichter SB, Quattrin T, Russell WE, Sunil B, Willi SM, Knecht LA, Niemoeller E, Licaj I, Schmider W, Miller D, DiMeglio LA. Safety and pharmacokinetics of teplizumab in children less than 8 years of age with stage 2 type 1 diabetes. Diabetologia. 2026 Feb;69(2):330-342. doi: 10.1007/s00125-025-06586-1. Epub 2025 Nov 6. PMID 41196293
- [Derived] Novograd J, Frishman WH. Teplizumab Therapy to Delay the Onset of Type 1 Diabetes. Cardiol Rev. 2024 Nov-Dec 01;32(6):572-576. doi: 10.1097/CRD.0000000000000563. Epub 2023 May 9. PMID 37158990